CLINICAL TRIAL: NCT06248229
Title: A Single Center, Flexible-Dose, 10-Week, Randomized, Double-Blinded, Placebo-Controlled, Clinical Trial To Study The Efficacy Of Dyanavel XR In Treating Co-Occurring Fatigue In Adults With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Trial of Dyanavel XR in Treating Co-occurring Fatigue Symptoms in Adults With Attention Deficit Hyperactivity Disorder (ADHD).
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rochester Center for Behavioral Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dyan24
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Fatigue; Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder
MeSH Terms: conditions — Fatigue; Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

STUDY DESIGN:
Intervention Model Description: 8-week single center, randomized, double-blind, placebo-controlled, flexible titration trial evaluating the efficacy of Dyanavel (Dyanavel XR) XR in the treatment of fatigue symptoms in adult subjects with a diagnosis of ADHD. Subjects will be randomly assigned (1:1) to a Dyanavel (Dyanavel XR) XR (flexible titration dosing) group (n = 22 to 25) or placebo group (n = 22 to 25). The study will utilize an intent to treat model and impute data, if statistically feasible, from dropouts utilizing a MNAR (missing not at random) approach.
  50 subjects qualifying for a ADHD diagnosis with co-occurring clinically significant fatigue symptoms will be randomized into the trial in two groups to ensure a minimum of 44 subjects completing the trial ( 25 per group, 10% hypothesized attrition rate).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the unblinded pharmacist will be aware of the subject's assigned group for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dyanavel XR (Active Agent) (Active Comparator): Dyanavel 5, 10, 15 or 20 mg once daily in the morning
  Interventions: Drug: Dyanavel XR
- Placebo (Placebo Comparator): Matching placebo 5, 10, 15 or 20 mg once daily in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dyanavel XR — Dosing will begin the morning following Visit 2. Subjects in the active group will begin the study on 5 mg of Dyanavel XR. Subjects will be advised to take one capsule each morning upon awakening, dosed consistently with respect to time. Subjects will be advised that tablets should be swallowed whole, not crushed, chewed, or cut. Subjects can take Dyanavel XR with or without food.
  Subjects will return to the study site on a weekly (and later, bi-weekly) basis for evaluation of symptoms and possible side effects. Subjects will be titrated to their optimal dose based on the dose titration schedule displayed in Section 5.1. The PI will be available to consult with patients as needed between Week 0 and Week 4 to adjust dosage per the PI's clinical judgment.
  Arms: Dyanavel XR (Active Agent)
Drug: Placebo — Dosing will begin the morning following Visit 2. Subjects in the placebo group will begin the study on 5 mg of placebo. Subjects will be advised to take one tablet each morning upon awakening, dosed consistently with respect to time. Subjects will be advised that tablets should be swallowed whole, not crushed, chewed, or cut. Subjects can take Dyanavel XR with or without food.
  Subjects will return to the study site on a weekly (and later, bi-weekly) basis for evaluation of symptoms and possible side effects. Subjects will be titrated to their optimal dose based on the dose titration schedule displayed in Section 5.1. The PI will be available to consult with patients as needed between Week 0 and Week 4 to adjust dosage per the PI's clinical judgment.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to study the impact of Dyanavel on co-occuring fatigue in adults with Attention Deficit/Hyperactivity Disorder. The main question it aims to answer is whether Dyanavel XR leads to a statistically significant reduction in fatigue compared to placebo, as measured by the Fatigue Symptom Inventory.

DETAILED DESCRIPTION:
10-week single center, randomized, double-blind, placebo-controlled, flexible titration trial evaluating the efficacy of Dyanavel (Dyanavel XR) XR in the treatment of fatigue symptoms in adult subjects with a diagnosis of ADHD. Subjects will be randomly assigned (1:1) to a Dyanavel (Dyanavel XR) XR (flexible titration dosing) group (n = 22 to 25) or placebo group (n = 22 to 25). The study will utilize an intent to treat model and impute data, if statistically feasible, from dropouts utilizing a MNAR (missing not at random) approach.

ELIGIBILITY:
Inclusion Criteria:

* At screening, all subjects must have a Fatigue Symptom Inventory average score on both of the interference and severity scales greater than 3.
* At screening, all subjects must score in the clinically significant range on the ADHD-RS-IV, meaning a score greater than 36.
* At screening, all subjects must meet criteria for an ADHD diagnosis as determined by the SCID-5 ADHD module.
* All subjects must be 18-65 years of age at the time of consent.
* All sexually active males or females of child baring potential must agree to practice two different methods of birth control or remain abstinent during the course of the trial. Methods of birth control or contraception will be logged. Male and female contraception will be continued throughout the study and for 30 days after study discontinuation. Women of childbearing potential must test negative for pregnancy at the Screening Visit.
* All subjects must live within the state of Michigan during the duration of the trial or be able to commute to the study site from a neighboring state with no more than a 50 mile one-way driving distance.
* All subjects must be able to swallow intact tablets.
* Subjects, in the opinion of the investigator, must be able to understand and comply with protocol requirements- including assessments, prescribed dosage regimens, and discontinuation of concomitant medications.
* All subjects must have a minimum level of intellectual functioning without evidence of significant general intellectual deficit, as determined by the primary investigator. Specific learning disorders will not be considered general intellectual deficits.
* All subjects must be able to provide written, personally signed and dated informed consent to participate in the study in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations before completing any study related procedures.
* All subjects must be fluent in English and have a degree of understanding sufficient to communicate suitably with the primary investigator and the study coordinator.
* Subjects must have a negative drug screen for methamphetamine, cocaine and other illicit drugs (illegal for recreational use in the State of Michigan) excluding cannabis due to legality of cannabis in Michigan. Subjects with a positive drug screen for confirmed prescription or over the counter use of medications will require the necessary washout per PI instruction. Subjects who test positive for any prohibited medications per PI may be permitted with PI approval. Re-tests will not be allowed for a positive screen of an illicit drug.
* All subjects must score at or above a 4 on the CGI-S at screening

Exclusion Criteria:

* Subjects must not be an immediate family of the Investigator or others directly affiliated with the study.
* Subjects must not have received treatment with a drug that has not received regulatory approval or participated in a clinical trial within 30 days prior to screening.
* Subjects must not have medical complications arising from being severely underweight or overweight.
* Subjects must not have a current comorbid psychiatric disorder that is uncontrolled and associated with significant symptoms or that requires a prohibited medication or behavioral modification program. Comorbid psychiatric diagnoses will be assessed during a psychiatric intake and scoring of the SCID and MINI. The Investigator will review on a case by case basis.
* Subjects must not currently be considered a suicide risk (as determined by the primary investigator and assessed by the C-SSRS). They must not have made a suicide attempt within the past two years. They cannot have current suicidal ideation with intent and plan to act, or current suicidal behavior.
* Subjects must not have a history of substance abuse or drug dependence according to DSM-5 criteria currently or within one year prior to study participation, excluding nicotine and caffeine. This is determined through clinical history and symptom checklist to be obtained at visit 1.
* Subjects must not test positive for an illicit substance at the time of screening.
* Subjects must not have a serious chronic or acute unstable medical condition or illness, including cardiovascular, renal, hepatic, respiratory, or hematologic illness, narrow angle glaucoma, or other unstable medical or psychiatric conditions that in the opinion of the Investigator would compromise participation or would likely lead to hospitalization during the duration of the study. Subjects with a history of intellectual impairment or a severe learning disability are also excluded.
* Subjects must not have a history of seizure disorder (other than infantile febrile seizures), any tic disorder, current diagnosis and/or family history of Tourette's disorder.
* Subjects must not have a history of organic heart disease including coronary artery disease, past myocardial infarction, angina, arrhythmias, congestive heart failure, valvular heart disease and congenital heart disease.
* Subjects must not be likely (as assessed by the primary investigator) to add psychotropic medications, apart from their current regimen or the drug under study, to their treatment regimen during the course of the study.
* Subjects must not have been previously enrolled in this study.
* Subjects must not anticipate relocation outside the geographic range of the investigative site during participation in the study. Subjects must not have extended travel plans inconsistent with the recommended visit intervals.
* Subjects must not be taking any excluded medications that cannot be discontinued prior to beginning treatment with study medication. Subjects' medical history will be reviewed by the PI and current prescription regimen will be reviewed for wakefulness-promoting drugs including CNS stimulants, histaminergic, noradrenergic and dopaminergic medications, as well as CYP2D6 inhibitors. The primary investigator will determine on a case by case basis if concomitant use of the patient's current prescriptions would affect response to Dyanavel XR. Stimulant medications must be washed out prior to baseline (methylphenidate or amphetamine based).
* Subjects must not have a known hypersensitivity, allergy intolerance or documented history of non-responsivity to amphetamine-based medications.
* Subjects who, in the opinion of the Investigator, are unsuitable in any other way to participate in the study.
* Subjects who have taken an MAOI within 14 days of the beginning of the study.
* Subjects currently taking a medication regimen that would otherwise likely interfere with the efficacy of Dyanavel XR or the integrity of study results as determined on a case by case basis by the primary investigator.
* Subjects who have recently (within the previous 3 months) been on CNS stimulant medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Symptom Inventory (FSI) | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Rating scale completed by study coordinator or PI. Score would be 0-10 with 10 being a worse outcome.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Functioning- Adult (BRIEF-A) | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Rating scale to assess subject's cognitive functioning. T scores are used to interpret the individual's level of executive functioning, and are derived from their raw scores. T-scores of 65 or over are considered clinically significant.
ADHD Rating Scale (ADHD-RS) | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Rating scale to evaluate symptoms of adult ADHD. Scores range from 0-54, with higher scores indicates a worse outcome.
ADHD Quality of Life Scale (ADHDQOL) | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Rating scale to assess quality of life, with possible scores ranging from 0-100. Higher scores are indicative of a better outcome.
Clinical Global Impression Scales (CGI) | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Clinician's subjective rating of subject's severity on a 7-point likert scale from 0-7, with higher scores indicative of a worse outcome.
Epworth Sleepiness Scale (ESS) | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Rating scale to assess level of daytime sleepiness. Scoers range from 0-24 with higher scores indicative of a worse outcome.
Insomnia Severity Index (ISI) | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Rating scale to assess level of insomnia. Scores range from 0-28 with higher scores indicative of a worse outcome.
Fibromyalgia Impact Questionnaire | Screening, Baseline, weeks 1, 2, 3, 4, 6 and 8
  Rating scale to assess subject's symptoms of fibromyalgia. Scores can range from 0-80, with higher scores indicative of a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Young, MD, Principal Investigator — Medical Director
Locations (1):
- Rochester Center for Behavioral Medicine, Rochester Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No